CLINICAL TRIAL: NCT00824161
Title: A Phase II Study of TAS-109 Given by Continuous Intravenous 14-day Infusion in Patients With Chemotherapy-refractory Advanced Colorectal Cancer
Brief Title: Phase II Study of TAS-109 to Treat Advanced Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAS109-0403
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Advanced Colorectal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): TAS-109
  Interventions: Drug: TAS-109

INTERVENTIONS:
Drug: TAS-109 — 14-day continuous central intravenous infusion at a dose of 2.0 mg/m2/day followed by a 7-day rest period.
  Number of cycles: until unacceptable toxicity or disease progression requires discontinuation.

SUMMARY:
The purpose of this study is to evaluate progression free survival primarily. The secondary objectives are to evaluate the antitumor activity, as assessed by objective tumor response, duration of clinical benefit, overall survival, and the safety profile of TAS-109

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal adenocarcinoma
* Received prior therapy, at least two regimens, containing a fluoropyrimidine, oxaliplatin, and irinotecan
* Have at least one measurable tumor, as defined by RECIST
* Must be capable of maintaining a central venous line access

Exclusion Criteria:

* Had previous anti-tumor therapy in the 3 weeks prior to study entry
* Have not recovered from all toxicities (excluding alopecia) from prior therapy to baseline or ≤grade 1 prior to study entry
* Have another malignancy in the past 3 years except curatively treated non-melanoma skin cancer or carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Xiong, M.D., Ph.D., Principal Investigator — The Center for Cancer and Blood Disorders
Locations (3):
- United States (3):
  - NYU Cancer Institute, East 34th Street, New York, New York
  - The University of Texas M.D. Anderson Cancer Center, Holcombe Boulevard, Houston, Texas
  - The Center for Cancer and Blood Disorders, West Magnolia Avenue, Fort Worth, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with chemotherapy-refractory advanced colorectal cancer have been recruited at 3 study sites in US between January 2009 and November 2009.
Pre-assignment Details: No screening period.
Groups:
- TAS-109: TAS-109 2.0 mg/m^2/day
Period: Overall Study
Arm/Group | TAS-109
Started | 28
Completed | 26
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Screen Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | TAS-109
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 55.8 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Progression Free Survival
Description: The primary endpoint was percentage of progression free survival as defined by the percentage of patients without progressive disease(PD)or death, whichever came first, at 3 months of therapy.
Time Frame: From date of randomization until date of the first documented progressive disease (PD) or death from any cause, whichever came first, assessed up to 3 months.
Population: Analysis was Intent to treatment(ITT) population.
Measure: Number (95% Confidence Interval); unit: percentage of PFS patients
Groups:
- TAS-109: TAS-109 2.0 mg/m^2/day Independent Assessment
Arm/Group | TAS-109
Number analyzed (Participants) | 28
percentage of PFS patients | 75.0 [55.1 to 89.3]

2. Secondary Outcome: Antitumor Activity
Description: Per RECIST Criteria and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall response rate was defined as percentage of patients of CR plus PR in ITT population.
Time Frame: From the date of initial treatment until the date of the first objective documentation of PD or death from any cause.
Population: Intent to treatment(ITT)
Measure: Number (95% Confidence Interval); unit: percentage of CR plus PR patients
Arm/Group | TAS-109
Number analyzed (Participants) | 28
percentage of CR plus PR patients | 0 (0) [0.0 to 12.3]

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the period from the date of first dose of TAS-109 to death date.
Time Frame: From the initial treatment until 12 months after enrollment of the last patient.
Population: Analysis was Intent to Treat(ITT) population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAS-109
Number analyzed (Participants) | 28
months | 5.5 [3.7 to NA] — As this study was terminated on the way, the upper bound of 95% CI was not calculated.

ADVERSE EVENTS:
Time Frame: Patients were monitored for any adverse events from the time of signed Informed Consent Form through 30 days post study medication.
Arm/Group | TAS-109
Serious Adverse Events (participants affected / at risk) | 9/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAS-109 (N=26)
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Disease progression (General disorders) | 2
Pyrexia (General disorders) | 1
Catheter bacteremia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAS-109 (N=26)
Anaemia (Blood and lymphatic system disorders) | 7
Leukopenia (Blood and lymphatic system disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Tachycardia (Cardiac disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 4
Ascites (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 10
Proctalgia (Gastrointestinal disorders) | 2
Small Intestinal Obstruction (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 7
Chills (General disorders) | 3
Disease Progression (General disorders) | 2
Fatigue (General disorders) | 14
Oedema Peripheral (General disorders) | 2
Pyrexia (General disorders) | 4
Hepatomegaly (Hepatobiliary disorders) | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Jaundice (Hepatobiliary disorders) | 2
Pneumonia (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 3
Blood Alkaline Phosphatase Increased (Investigations) | 3
Haemoglobin Decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 2
Dysuria (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 6
Deep Vein Thrombosis (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No